CLINICAL TRIAL: NCT01850394
Title: Efficacy of Low-dose Intra-articular Tranexamic Acid in Total Knee Replacement; A Prospective Triple-blinded Randomized Controlled Trial.
Brief Title: Efficacy of Low-dose Intra-articular Tranexamic Acid in Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Viroj Kawinwonggowit, Clinical Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID 01-53-06
Record Dates: First submitted 2013-05-02; First posted 2013-05-09 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Primary Osteoarthritis of Knee Nos
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Placebo Comparator): physiologic saline 25 ml
  Interventions: Drug: Physiologic saline
- TXA-250 group (Active Comparator): A total of 25-ml solution with 250-mg tranexamic acid
  Interventions: Drug: Tranexamic Acid; Drug: Physiologic saline
- TXA-500 group (Active Comparator): A total of 25-ml solution with 500-mg tranexamic acid
  Interventions: Drug: Tranexamic Acid; Drug: Physiologic saline

INTERVENTIONS:
Drug: Tranexamic Acid — Inject tranexamic acid solution intra-articularly after fascia closure
  Other Names: Transmin
  Arms: TXA-250 group; TXA-500 group
Drug: Physiologic saline — Use physiologic saline for mixing with tranexamic acid or use alone in placebo group

SUMMARY:
The purpose of this study is to determine 1) the effective dosage of intra-articular tranexamic acid injection for controlling blood loss and blood transfusion requirement in conventional total knee replacement, and 2) whether the blood loss reduction effect depended on the dose of tranexamic acid used.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as primary knee osteoarthritis and underwent unilateral primary cemented conventional total knee replacement
* no risk of abnormal bleeding tendency or bleeding disorder (normal coagulogram, serum creatinine < 2.0 mg/dL, stop nonsteroidal anti-inflammatory drugs and antiplatelet drugs more than 7 days
* no contra-indication for tranexamic acid use (no active intravascular clotting process, no acquired defective colour vision, no subarachnoid hemorrhage, no hypersensitivity to TXA, and no any of history of serious adverse effects, thrombotic disorder and hematuria)

Exclusion Criteria:

* incomplete data collection, for example, malfunctioned drain or accidental drain removal.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Sa-Ngasoongsong P, Channoom T, Kawinwonggowit V, Woratanarat P, Chanplakorn P, Wibulpolprasert B, Wongsak S, Udomsubpayakul U, Wechmongkolgorn S, Lekpittaya N. Postoperative blood loss reduction in computer-assisted surgery total knee replacement by low dose intra-articular tranexamic acid injection together with 2-hour clamp drain: a prospective triple-blinded randomized controlled trial. Orthop Rev (Pavia). 2011;3(2):e12. doi: 10.4081/or.2011.e12. Epub 2011 Jun 29. PMID 22053253
- [Background] Ishida K, Tsumura N, Kitagawa A, Hamamura S, Fukuda K, Dogaki Y, Kubo S, Matsumoto T, Matsushita T, Chin T, Iguchi T, Kurosaka M, Kuroda R. Intra-articular injection of tranexamic acid reduces not only blood loss but also knee joint swelling after total knee arthroplasty. Int Orthop. 2011 Nov;35(11):1639-45. doi: 10.1007/s00264-010-1205-3. Epub 2011 Jan 21. PMID 21253725
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Maniar RN, Kumar G, Singhi T, Nayak RM, Maniar PR. Most effective regimen of tranexamic acid in knee arthroplasty: a prospective randomized controlled study in 240 patients. Clin Orthop Relat Res. 2012 Sep;470(9):2605-12. doi: 10.1007/s11999-012-2310-y. Epub 2012 Mar 15. PMID 22419350
- [Background] Roy SP, Tanki UF, Dutta A, Jain SK, Nagi ON. Efficacy of intra-articular tranexamic acid in blood loss reduction following primary unilateral total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2494-501. doi: 10.1007/s00167-012-1942-5. Epub 2012 Mar 15. PMID 22419263
- [Background] Seo JG, Moon YW, Park SH, Kim SM, Ko KR. The comparative efficacies of intra-articular and IV tranexamic acid for reducing blood loss during total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2013 Aug;21(8):1869-74. doi: 10.1007/s00167-012-2079-2. Epub 2012 Jun 24. PMID 22729012
- [Derived] Sa-Ngasoongsong P, Wongsak S, Chanplakorn P, Woratanarat P, Wechmongkolgorn S, Wibulpolprasert B, Mulpruek P, Kawinwonggowit V. Efficacy of low-dose intra-articular tranexamic acid in total knee replacement; a prospective triple-blinded randomized controlled trial. BMC Musculoskelet Disord. 2013 Dec 5;14:340. doi: 10.1186/1471-2474-14-340. PMID 24308672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients, who planned to undergo primary total knee replacement, were recruited from medical clinics before setting the operative schedule between 2009 and 2010.
Pre-assignment Details: Seventeen patients were excluded that including refusal to participate (4 patients), serum creatinine more than 2.0 mg% (4 patients), rheumatoid arthritis (4 patients), abnormal coagulogram (3 patients), and history of stroke (2 patients)
Groups:
- Control Group: physiologic saline 25 ml
  Physiologic saline : Use physiologic saline for mixing with tranexamic acid or use alone in placebo group
- TXA-250 Group: A total of 25-ml solution with 250-mg tranexamic acid
  Physiologic saline : Use physiologic saline for mixing with tranexamic acid or use alone in placebo group
  Tranexamic Acid : Inject tranexamic acid solution intra-articularly after fascia closure
- TXA-500 Group: A total of 25-ml solution with 500-mg tranexamic acid
  Physiologic saline : Use physiologic saline for mixing with tranexamic acid or use alone in placebo group
  Tranexamic Acid : Inject tranexamic acid solution intra-articularly after fascia closure
Period: Overall Study
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Started | 45 | 45 | 45
Completed | 45 | 45 | 45
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group | Total
Number analyzed (Participants) | 45 | 45 | 45 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 13 | 53
  >=65 years | 25 | 25 | 32 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.3) | 67.6 (8.7) | 68.1 (6.2) | 67.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 40 | 125
  Male | 2 | 3 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Thailand | 45 | 45 | 45 | 135

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Blood Loss
Description: * Drainage blood loss measured by accumulating total drainage volume postoperatively
  * Calculated total blood loss measured by using specific formula and difference between hematocrit preoperatively and the fourth postoperative day
Time Frame: 5 days after surgery
Population: Using intention-to-treat analysis
Measure: Median (Standard Deviation); unit: ml
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Number analyzed (Participants) | 45 | 45 | 45
ml
  Drainage blood loss | 546.9 (273.0) | 475.0 (254.4) | 430.2 (224.0)
  Calculated total blood loss | 329.2 (119.4) | 239.7 (83.7) | 217.2 (86.1)
Statistical Analysis 1: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 180, Standard Deviation 300
Statistical Analysis 2: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Net) = 150, Standard Deviation 200

2. Secondary Outcome: Knee Function Scores
Description: Knee function score was measured with 2 methods, and were evaluated preoperatively and then postoperatively at 3-month, 6-month, and 1-year period.
  1. Knee Society Knee Score using for rating knee function measurement and subdivided into two parts; knee score and function score 1.1. Knee score : calculated from pain, presence of deformity, total range of flexion, alignment, and stability. Total score is 100 (0-100), more score means better.
     1.2. Function score : calculated from patient's ability to walk and climb stairs. The score ranges from 0-100, more score means better.
  2. Western Ontario and McMaster Universities Arthritis Index or WOMAC score : a widely used, standardized questionnaires for evaluating the condition of patients with knee osteoarthritis, including pain (score = 0-20), stiffness (0-8), and functional limitation (0-68). Total score ranges from 0-68, lower score means better.
Time Frame: 1 year after surgery
Population: Using intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Number analyzed (Participants) | 45 | 45 | 45
units on a scale
  Knee Society Knee score at 1 year | 148.9 (10.1) | 151.2 (9.1) | 150.9 (9.3)
  WOMAC score at 1 year | 15.5 (6.6) | 15.1 (6.2) | 14.5 (7.1)
Statistical Analysis 1: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 140, Standard Deviation 15
Statistical Analysis 2: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, ANOVA; Mean Difference (Final Values) = 15, Standard Deviation 4

3. Secondary Outcome: Number of Patients Required Blood Transfusion
Time Frame: postoperative period (5 days after surgery)
Measure: Number; unit: participants
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Number analyzed (Participants) | 45 | 45 | 45
participants | 10 | 6 | 0
Statistical Analysis 1: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, Fisher Exact; Hazard Ratio (HR) = 0.25, Standard Error of Mean 0.1

4. Secondary Outcome: Number of Patients Having Postoperative Complications
Description: Postoperative complications were measured as an incidence of the following complications;
  * wound hematoma
  * surgical site infection
  * systemic infection
  * deep vein thrombosis
  * pulmonary embolism
  * knee stiffness requiring manipulation
  * medical complication such as myocardial infarction, congestive hear failure
Time Frame: postoperative 1-year period
Population: Using Intention-to-treat analysis
Measure: Number; unit: participants
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Number analyzed (Participants) | 45 | 45 | 45
participants
  Re-clamp incidence | 6 | 1 | 0
  Re-dressing incidence | 3 | 0 | 0
  Venous thromboembolic complication | 4 | 1 | 2
  Congestive heart failure | 0 | 1 | 0
Statistical Analysis 1: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p < 0.05, Fisher Exact; Hazard Ratio (HR) = 0.1, Standard Error of Mean 0.02

5. Primary Outcome: Total Hemoglobin Loss
Description: Total hemoglobin loos measured by difference between hemoglobin preoperatively and the fourth postoperative day
Time Frame: 5 days after surgery
Population: Use intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Number analyzed (Participants) | 45 | 45 | 45
g/dL | 2.9 (1.2) | 2.2 (0.7) | 2.2 (0.7)
Statistical Analysis 1: Comparison: Control Group vs TXA-250 Group vs TXA-500 Group; Test type: Superiority or Other; p = 0.05, ANOVA; Mean Difference (Net) = 0.66, Standard Deviation 1.0

ADVERSE EVENTS:
Time Frame: 5 days
Description: Perioperative venous thromboembolic complications
  * deep vein thrombosis screened with duplex doppler ultrasound in all cases
  * pulmonary embolism diagnosed with clinical hypoxemia and confirmed with computer tomography angiogram
Arm/Group | Control Group | TXA-250 Group | TXA-500 Group
Serious Adverse Events (participants affected / at risk) | 4/45 | 1/45 | 2/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=45) | TXA-250 Group (N=45) | TXA-500 Group (N=45)
Venous thromboembolic complication (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No